CLINICAL TRIAL: NCT05245786
Title: Pilot Study: Imaging Tumor Extent and Response Before and After Neoadjuvant Chemotherapy and Radiotherapy in Locally Advanced Rectal Cancer Using 64Cu-Labeled M5A Antibody to Carcinoembryonic Antigen (CEA)
Brief Title: An Investigational Scan (64Cu-Labeled M5A Antibody) in Combination With SOC Chemotherapy and Radiotherapy in Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20439; NCI-2021-14005 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20439 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-01-11; First posted 2022-02-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Rectal Carcinoma; Stage III Rectal Cancer AJCC v8; Stage IIIA Rectal Cancer AJCC v8; Stage IIIB Rectal Cancer AJCC v8; Stage IIIC Rectal Cancer AJCC v8
MeSH Terms: conditions — Rectal Neoplasms | interventions — Copper; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (64Cu labeled M5A antibody and imaging) (Experimental): Patients receive 64Cu labeled M5A antibody IV over 5 minutes on day 0 pre standard of care chemo/radiotherapy and on day 0 post chemo/radiotherapy. Patients also undergo 64Cu-M5A PET scan on day 1 pre chemo/radiotherapy and on day 1 post chemo/radiotherapy.
  Interventions: Biological: Copper Cu 64 Anti-CEA Monoclonal Antibody M5A; Procedure: Imaging Technique

INTERVENTIONS:
Biological: Copper Cu 64 Anti-CEA Monoclonal Antibody M5A — Given IV
  Other Names: 64Cu-DOTA-M5A; Cu 64-M5A
Procedure: Imaging Technique — Undergo imaging
  Other Names: Diagnostic Imaging Technique; Imaging; imaging procedure; Imaging Procedures; imaging type; imaging_type; Medical Imaging; Type of imaging

SUMMARY:
This early phase I trial investigates how well 64Cu-labeled M5A antibody scan works in assessing tumor activity before and after patients with rectal cancer that has spread to nearby tissue or lymph nodes (locally advanced) who are undergoing chemotherapy and radiotherapy. Using 64Cu-labeled M5A positron emission tomography imaging may play a significant role in imaging patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the Copper Cu 64 anti-carcinoembryonic antigen (CEA) monoclonal antibody M5A (64Cu labeled M5A antibody) demonstrates a potentially impactful finding for patient management either in the pre-treatment scan (potentially impacting choice of therapy or impacting the radiotherapy [RT] plan) or the scan immediately prior to planned surgery (after standard care [SOC] chemoradiation) in patients with locally advanced rectal cancer.

SECONDARY OBJECTIVES:

I. To determine the safety of administration of 64Cu labeled M5A antibody. II. To describe/summarize each of the 15 patients' 64Cu-M5A positron emission tomography (PET) imaging findings and corresponding SOC scans and pathology.

OUTLINE:

Patients receive 64Cu labeled M5A antibody intravenously (IV) over 5 minutes on day 0 pre standard of care chemo/radiotherapy and on day 0 post chemo/radiotherapy. Patients also undergo 64Cu-M5A PET scan on day 1 pre chemo/radiotherapy and on day 1 post chemo/radiotherapy.

After completion of the study treatment, patients medical records are reviewed up to 2-3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed CEA expressing locally advanced rectal cancer (T3, T4 and N0 or N plus [+])
* Patients must be 18 years of age or older
* The effects of 64Cu-M5A on the developing fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence} prior to study entry and for six months following duration of study participation. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Patients must have a known site of disease. Patients must be scheduled to undergo neoadjuvant chemotherapy and radiation therapy followed by surgery
* Patients who are planned for total neoadjuvant therapy where additional chemotherapy is planned before neoadjuvant chemoradiotherapy (CRT) are also eligible
* Although not mandated by the protocol, the results of the computed tomography (CT), magnetic resonance imaging (MRI) and fludeoxyglucose F-18 (FDG) PET scans and labs (blood cell count [CBC], comprehensive metabolic panel [CMP]) that are performed as part of the standard work up should be available and should have been done within 2 months prior to study entry
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Prior therapy (chemotherapy, immunotherapy, radiotherapy) must be completed at least 2 weeks prior to infusion of radiolabeled antibody

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection
* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 64Cu-M5A
* Pregnant women are excluded from this study because 64Cu-M5A is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ^64Cu-M5A, breastfeeding should be discontinued if the mother is treated with 64Cu-M5A
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2026-11-12 (Estimated); Study Completion 2026-11-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with impactful finding using 64Cu-M5A positron emission tomography (PET) imaging. | Up to 3 years
  We seek to evaluate the potential for 64Cu-M5A PET imaging in locally advanced rectal cancer before and after neoadjuvant radio-chemotherapy yet prior to planned surgery. Scan findings will be compared to standard of care imaging studies (eg. CT, MRI and FDG PET scans) and biopsy and findings from endoscopy and surgery performed post neoadjuvant CRT therapy. Each of the 15 cases will be reviewed in a protocol team meeting consisting of a radiologist, radiation oncologist, surgeon and pathologist. Cases will be determined by consensus. Examples of "potentially impactful" would be 1) any new lesion not seen on other imaging modalities and confirmed by pathology, 2) a negative 64CuM5A PET on a suspicious lesion by standard of care (SOC) determined to be negative on pathology, or 3) other important differences as judged by the evaluation team including if findings from initial 64CuDOTA-M5A immunoPET imaging could result in modification and adaption of the radiotherapy plan.

SECONDARY OUTCOMES:
Count of Adverse Events. | Up to 3 years
  The frequency and severity of any adverse events possibly related to 64Cu-M5A PET.
  The toxicity will be graded using the NCI common toxicity scale CTCAE v 5.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Y Wong, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States